CLINICAL TRIAL: NCT05188287
Title: Identifying the Barriers and Facilitators of Participation in mHealth Research Among African Americans Using a Mixed-Methods Approach.
Brief Title: A Culturally Tailored Smartphone Application for African American Smokers
Acronym: HC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14094; K01MD015295 (NIH)
Record Dates: First submitted 2021-12-26; First posted 2022-01-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HealthyCells (Experimental): The HealthyCells app will have the following features:
  Smoking status assessments with facial recognition: Participants will initiate a smoking status assessment and CO breath sample submission using the iCOquit® Smokerlyzer® TWICE per day. To verify the participant's identity while they complete their CO breath sample, we will use Microsoft Face API.
  Daily step counter and sedentary behavior prompts: A Google OS smartwatch will be used to monitor participants' activity, and the HealthyCells app will deliver an activity prompt when they have been sedentary for 30 minutes, which will be experienced as noise and vibration on the phone and watch. Also, a text-based reminder message will appear on the phone and watch along with a "personalized tip" for reducing sedentary time.
  Motivational messages for smoking cessation and physical activity. TWICE per day, the HealthyCells app will send messages to encourage users to remain quit and become more active.
  Interventions: Behavioral: HealthyCells

INTERVENTIONS:
Behavioral: HealthyCells — Smoking cessation smartphone app

SUMMARY:
The overall objectives of this research proposal, are to (a) create a smartphone application for smoking cessation (i.e., HealthyCells), which will be achieved by integrating two pre-existing evidence-based smartphone interventions, (b) create culturally tailored treatment content (i.e., messages, images, and videos) for African American smokers, and (c) evaluate the feasibility of HealthyCells at addressing smoking and sedentary behavior among African Americans. A pilot sample of African American smokers (N = 15) will briefly use the HealthyCells app and provide critical feedback through semi-structured interviews to refine the smartphone intervention. Once the HealthyCells app is refined, African Americans (N = 30) who are interested in quitting smoking will use the app during a scheduled quit attempt. Starting on the scheduled quit date, HealthyCells will prompt participants to complete twice-daily remote smoking status assessments to earn rewards for abstinence. The app will deliver real-time messages telling participants to stand up and move around during prolonged bouts of sedentary behavior (i.e., ≥ 30 minutes of uninterrupted time spent in a sitting, reclining, or lying posture). Participants will also have on-demand access to culturally tailored information and strategies for remaining abstinent and reducing sedentary behavior within the HealthyCells app. The primary outcomes will be biochemically confirmed point prevalence smoking abstinence at 8 weeks post-quit date, and the difference in sedentary time 7 consecutive days before quitting compared with 7 consecutive days at 8-weeks post-quit, as measured by a research-grade accelerometer.

DETAILED DESCRIPTION:
African Americans are interested in quitting smoking, they attempt to quit smoking at a higher rate than Whites, yet they have lower cessation rates compared to Whites and many other racial/ethnic groups. Successfully increasing cessation rates among African Americans would reduce the racial disparity in mortality between African Americans and Whites by up to 20%. Many smoking cessation interventions include physical activity components to boost cessation rates, but no studies have attempted to promote sedentary behavior reduction as a cessation strategy, which may plausibly share similar benefits with physical activity, such as increased self-efficacy for smoking cessation and reduced smoking urges and cravings.

African Americans also face numerous barriers to seeking in-person treatment for smoking cessation, and research has shown that the use of smartphones can facilitate intensive behavioral interventions without requiring burdensome in-person treatment. Smartphone interventions can also be tailored to address the specific needs of African Americans (e.g., discrimination, and financial strain), and capitalize on cultural strengths (e.g., spirituality and collectivism) to reduce barriers and encourage behavior change. The research team has developed numerous evidence-based smartphone interventions to address a range of modifiable health risk factors among vulnerable populations, which are capable of being culturally tailored for African Americans. One intervention is a smartphone-based contingency management intervention that provides financial rewards for smoking abstinence after remote verification of smoking status using low-cost portable carbon monoxide monitors and facial recognition software (i.e., PrevailGO). The other is a smartphone-based sedentary behavior reduction intervention that uses wrist-worn activity monitors in combination with smartphone technology to monitor activity in real-time and deliver activity prompts when individuals are engaged in prolonged bouts of sedentary behavior (i.e., SMARTpath). SMARTpath also provides graphical feedback about sedentary time over the past day, week, and month. Integrating and tailoring these evidence-based smartphone interventions for African Americans may equip them with the tools, skills, and information needed to remain abstinent from smoking.

The long-term goal of this research study is to improve smoking cessation outcomes among African Americans using evidence-based, culturally tailored smartphone interventions. The overall objectives of this research proposal, which is the next step toward achieving this long-term goal, are to (a) create a smartphone application for smoking cessation (i.e., HealthyCells), which will be achieved by integrating two pre-existing evidence-based smartphone interventions, PrevailGO and SMARTpath, (b) create culturally tailored treatment content (i.e., messages, images, and videos) for African American smokers for the HealthyCells app, and (c) evaluate the feasibility of HealthyCells at addressing smoking and sedentary behavior among African Americans. A pilot sample of African American smokers (N = 15) will briefly use the HealthyCells app and provide critical feedback through semi-structured interviews to refine the smartphone intervention. Once the HealthyCells app is refined, African Americans (N = 30) who are interested in quitting smoking will use the app during a scheduled quit attempt. Starting on the scheduled quit date, HealthyCells will prompt participants to complete twice-daily remote smoking status assessments to earn rewards for abstinence. The app will deliver real-time messages telling participants to stand up and move around during prolonged bouts of sedentary behavior (i.e., ≥ 30 minutes of uninterrupted time spent in a sitting, reclining, or lying posture). Participants will also have on-demand access to culturally tailored information and strategies for remaining abstinent and reducing sedentary behavior within the HealthyCells app. The primary outcomes will be biochemically confirmed point prevalence smoking abstinence (PPA) at 8 weeks post-quit date, and the difference in sedentary time 7 consecutive days before quitting compared with 7 consecutive days at 8-weeks post-quit, as measured by a research-grade accelerometer. The aims of this project are the following:

AIM 1: Create HealthyCells and populate the app with culturally tailored content for smoking cessation and sedentary behavior reduction. HealthyCells will be created by integrating PrevailGO with SMARTpath. Culturally tailored treatment content for smoking cessation and sedentary behavior reduction will be developed based on an extensive literature review. African American smokers (N = 15) will demo the HealthyCells application and participate in a post-demo semi-structured interview to obtain their overall impressions of the HealthyCells app and refine the culturally tailored treatment content.

AIM 2: Determine the feasibility and preliminary estimates of the effect of HealthyCells on smoking and sedentary behavior among African Americans. The primary objective is to determine whether the PPA prevalence and changes in sedentary time are sufficient to warrant further use of HealthyCells in this population (> 15% PPA at 8 weeks post-quit and > 30-minute daily net reduction in sedentary time). These feasibility thresholds are based on published findings from a smartphone-based contingency management intervention for smoking cessation and a smartphone-based sedentary behavior reduction intervention.

ELIGIBILITY:
Study Inclusion Criteria

* Must be 18 years of age or older
* Must identify as Black/African-American
* Must smoke at least 5 cigarettes or cigarette equivalents per day (i.e., cigarettes, cigars, and cigarillos)
* Must be willing to use NRT, a smartphone watch and app, and a smoking cessation counselor to help them quit smoking
* Must be willing to quit smoking within the next 3 weeks
* Must have a CO level of >6 ppm at app activation.
* Are not currently active, defined as engaging in less than 150 minutes of moderate-intensity aerobic physical activity (e.g., brisk walking) or 75 minutes of vigorous-intensity aerobic physical activity (e.g., running or jogging) each week?

Study Exclusion Criteria

* Does not give permission to administer screening survey
* Does not understand or speak English
* Is not a U.S. citizen or permanent U.S. resident
* Does not use tobacco products
* Does not want to provide SSN, residency status, or OUHSC employee status
* Is not willing to abstain from smoking marijuana or cannabis during their quit attempt
* Is not willing to upload a picture of their tobacco product
* Is not ready to quit smoking as defined by scoring 4 or lower on the readiness to quit ladder
* Has a medical condition that prevents the use of NRT without approval from a healthcare provider
* Has had a serious allergic reaction or side effect from the use of NRT
* Does not give permission to collect contact information
* Must not be currently active, defined as engaging in less than 150 minutes of moderate-intensity aerobic physical activity (e.g., brisk walking) or 75 minutes of vigorous-intensity aerobic physical activity (e.g., running or jogging) each week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically-Verified smoking cessation | 8 weeks
  Biochemically confirmed 7-day point prevalence abstinence using the CO criteria cutoff of ≤ 6 ppm
Accelerometer-verified reduction in sedentary time | 8 weeks
  Accelerometer-verified confirmation of a > 30-minute daily net reduction in sedentary time

CONTACTS AND LOCATIONS:
Overall Officials: Darla Kendzor, PhD, Study Chair — TSET Health Promotion Research Center
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide publicly archived de-identified datasets for all published papers related to the project so independent investigators can replicate our findings or use results for meta-analyses.
Supporting Information: Analytic Code
Time Frame: De-identified data will be made available one-year after the publication of the primary outcome data.
Access Criteria: Data can be requested from the primary study contact, or retrieved from public data repository.

REFERENCES:
- [Derived] Alexander A, Businelle M, Cheney M, Cohn A, McNeill L, Short K, Frank-Pearce S, Bradley D, Estrada K, Flores I, Fronheiser J, Kendzor D. An mHealth Intervention With Financial Incentives to Promote Smoking Cessation and Physical Activity Among Black Adults: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 31;14:e69771. doi: 10.2196/69771. PMID 39888657